CLINICAL TRIAL: NCT05538052
Title: Use of Tramadol Injections on the Anaesthetic Success Rate of Intraligamentary Injections in Patients With Symptomatic Irreversible Pulpitis
Brief Title: Use of Tramadol Intraligamentary Injections
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Jamia Millia Islamia (Other)
Responsible Party: Principal Investigator, Dr. Vivek Aggarwal, Professor, Jamia Millia Islamia
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 106
Record Dates: First submitted 2022-09-08; First posted 2022-09-13 (Actual); Last update posted 2022-12-19 (Actual); Status verified 2022-12

CONDITIONS: Pulpitis
MeSH Terms: conditions — Pulpitis | interventions — Tramadol; Lidocaine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Alpha-numeric codes
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- 2% lidocaine (Active Comparator): The first group will receive intraligamentary injections of 2% lidocaine with 1: 80 000 epinephrine. The injections will be administered using a pressure-type syringe (Osung Deosy, Pearland, Tx, USA) and 30 gauge short needles (Septojet needles, Septodont).
  Interventions: Drug: Lidocaine Hydrochloride
- 2% lidocaine plus tramadol hydrochloride (Experimental): The second group will receive intraligamentary injections of 2% lidocaine with 1:80 000 epinephrine plus tramadol hydrochloride (50 mg, 1:1 v/v ratio). The injections will be administered using a pressure-type syringe (Osung Deosy, Pearland, Tx, USA) and 30 gauge short needles (Septojet needles, Septodont).
  Interventions: Drug: Tramadol hydrochloride; Drug: Lidocaine Hydrochloride
- tramadol hydrochloride (Experimental): The second group will receive intraligamentary injections of tramadol hydrochloride (25mg/ mL). The injections will be administered using a pressure-type syringe (Osung Deosy, Pearland, Tx, USA) and 30 gauge short needles (Septojet needles, Septodont).
  Interventions: Drug: Tramadol hydrochloride

INTERVENTIONS:
Drug: Tramadol hydrochloride — Supplementary intraligamentary injections deposited in the gingival sulcus of the involved tooth
  Arms: 2% lidocaine plus tramadol hydrochloride; tramadol hydrochloride
Drug: Lidocaine Hydrochloride — Supplementary intraligamentary injections deposited in the gingival sulcus of the involved tooth
  Arms: 2% lidocaine; 2% lidocaine plus tramadol hydrochloride

SUMMARY:
Introduction: To achieve painless treatment in patients with a failed primary IANB, supplementary anaesthesia has been advised. The majority of the studies evaluating intraligamentary injections have been performed on asymptomatic teeth. Very limited research has been dedicated to the evaluation of different variables in intraligamentary injections in patients with symptomatic irreversible pulpitis Aim: To evaluate the anaesthetic efficacy of 2% lidocaine with 1:80 000 epinephrine vs. 2% lidocaine with 1:80 000 epinephrine plus tramadol hydrochloride (50 mg, 1:1 v/v ratio), given as intraligamentary injections after a failed inferior alveolar nerve block (IANB), in patients with symptomatic irreversible pulpitis. Objective: 1. To achieve painless treatment in patients with a failed primary IANB. during the endodontic management of symptomatic mandibular first/second molar. 2. To evaluate the heart rate during and after intraligamentary injections Methods: This prospective, randomized, double-blind clinical trial will be carried out by Conservative Dentistry, Faculty Of Dentistry, Jamia Millia Islamia. Sixty adult patients with symptomatic irreversible pulpits in a mandibular first or second molar will receive an initial IANB with 2% lidocaine with 1:80 000 epinephrine. Pain during the endodontic treatment will be assessed using a visual analogue scale(VAS). Patients experiencing pain on endodontic intervention shall be randomly allocated to one of the two treatment groups: one group shall receive 0.6 mL/ root of supplementary intraligamentary injection of 2% lidocaine with 1:80 000 epinephrine; while the second group shall receive 2% lidocaine with 1:80 000 epinephrine plus tramadol hydrochloride (50 mg, 1:1 v/v ratio). Endodontic treatment will be re-initiated. Success after primary injection or supplementary injection will be defined as no or mild pain (less than 55 mm on HP VAS) during access preparation and root canal instrumentation. Heart rate will be monitored using a finger pulse oximeter by a faculty member. Statistical analysis: The results will be tabulated in contingency tables. The anaesthetic success rates will be analyzed with the Pearson chi-square test at 5% significance levels. The heart rate changes will be analyzed using a t-test.

DETAILED DESCRIPTION:
Patients experiencing a failed primary IANB shall be enrolled in the study. The initial failure will be defined as pain (score more than 54 on Heft Parker Visual Analog Scale (VAS) during access cavity preparation or at the root canal instrumentation stage. The primary outcome (endpoint) will be defined as "success or failure, " indicating the ability to undertake pulp access and canal instrumentation with no or mild pain. The secondary outcome will be the evaluation of heart rate after supplementary intraligamentary injections.

A tentative sample size calculation has been performed using data from a previous study, keeping the α level type I error at 0.05 for a single-tailed test and β level type II error at 0.20.19 The analysis indicated that a sample size of 35 subjects would give 80% power to detect a 30% difference in the success rates of the two different supplemental intraligamentary injections. For heart rate analysis, it has been calculated that a minimum of 23 patients per group shall be required to detect a difference of 10 beats per minute (with a baseline heart rate of 72 beats per minute).

The treatment procedure and the use of pain scales will be explained to the patients. A combined VAS, the Heft-Parker scale (HP VAS), will be used in the present study.

All patients will receive a primary IANB injection using 1.8 mL of 2% lidocaine with 1: 80 000 epinephrine using a direct Halsted approach. The needle will be inserted until bony resistance will be felt. After reaching the target area, aspiration will be performed, and the solution will be deposited over a period of 60 seconds. After 10 minutes, the patients will be asked about lip numbness. Patients without profound lip numbness will be excluded from the study since the block will be considered 'missed'. A conventional access opening will be initiated after isolation with a rubber dam. Patients will be instructed to raise their hands if any pain will be felt during the procedure. In case of pain during treatment, the procedure will be stopped, and the patients will be asked to rate the pain on the HP VAS. The patients with failed primary IANB will receive supplementary intraligamentary injections of either 2% lidocaine with 1:80 000 epinephrine or 2% lidocaine with 1:80 000 epinephrine plus tramadol hydrochloride (50 mg, 1:1 v/v ratio) or tramadol hydrochloride (25mg/mL). The cartridges will be masked with an opaque tape and coded with an alpha-numeric code. The code will be broken only after the completion of the study. The patients will be randomly allocated to three treatment groups (n=105, 35 patients per group) with the help of an online random generator. The rubber dam will be removed and the injection site will be cleaned with an antiseptic solution. The resting heart rate will be monitored with a finger pulse oximeter by a faculty member. The first group will receive intraligamentary injections of 2% lidocaine with 1: 80 000 epinephrine. The injections will be administered using a pressure-type syringe (Osung Deosy, Pearland, Tx, USA) and 30 gauge short needles (Septojet needles, Septodont). The second group will receive intraligamentary injections of 2% lidocaine with 1:80 000 epinephrine plus tramadol hydrochloride (50 mg, 1:1 v/v ratio). The third group shall receive intraligamentary injections of tramadol hydrochloride (25mg/ mL). A total of 1.2 mL of anaesthetic solution will be deposited. The heart rate will be measured at 15-second intervals till 5 minutes after intraligamentary injections. Success will be again defined as no pain or faint/weak/mild pain during endodontic access preparation and instrumentation.

Statistical analysis: The results will be tabulated in contingency tables. The age of patients will be analyzed using the Mann-Whitney U test at P < .05. The gender and distribution of teeth will be analyzed using 2X2 contingency tables and chi-square tests. The anaesthetic success rates will be analyzed with the Pearson chi-square test. The heart rate changes will be analyzed using a t-test.

ELIGIBILITY:
Inclusion criteria:

1. Symptomatic carious exposed mandibular first or second molars.
2. Positive and prolonged response to thermal sensitivity tests and electric pulp test.
3. Vital coronal pulp on access cavity preparation.
4. American Society of Anesthesiologists class I or II medical history.
5. Ability to understand the use of pain scales.

Exclusion criteria

1. Active pain in more than 1 tooth.
2. Teeth with fused roots.
3. Radiographic evidence of an extra root.
4. Large restorations with overhanging margins.
5. Full crowns or deep periodontal pockets.
6. Known allergy or contraindications to any content of the local anaesthetic solution.
7. History of known or suspected drug abuse.
8. Taking any drugs which could affect the pain perception, e.g, opioids, antidepressants, anticonvulsants, muscle relaxants, anxiolytics, sedatives, NSAIDs. 23
9. Pregnant or breastfeeding patients.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 105 (Actual)
Dates: Start 2022-04-01 (Actual); Primary Completion 2022-11-30 (Actual); Study Completion 2022-11-30 (Actual)

PRIMARY OUTCOMES:
Anesthetic success rate | 15 minutes after the injections
  absence of any response to electric pulp testing and the ability of the clinician to perform endodontic access and root canal instrumentation with no or mild pain.

SECONDARY OUTCOMES:
Changes in heart rates | Immediately after the intraligamentary injections
  detection of any change in the heart rates after intraligamentary injections

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Dentistry, Jamia MIliia Islamia, New Delhi, India

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP